CLINICAL TRIAL: NCT05748470
Title: A Prospective, Single-center, Single-blind, Randomized Split-face Controlled Clinical Study to Evaluate the Efficacy and Satisfaction of Ultrasound Therapy Combined With SkinCeuticals A.G.E for Improving Facial Aging in Real World Clinical Practice
Brief Title: A Clinical Study to Evaluate the Efficacy and Satisfaction of Ultrasound Therapy Combined With SkinCeuticals A.G.E for Improving Facial Aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yes Skin Medical Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WSong
Record Dates: First submitted 2023-02-03; First posted 2023-02-28 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: SkinCeuticals A.G.E
- Control group (Active Comparator)
  Interventions: Other: standard cream

INTERVENTIONS:
Other: SkinCeuticals A.G.E — Ultrasound therapy combined with SkinCeuticals A.G.E + conventional moisturizing and sunscreen.
  Arms: Test group
Other: standard cream — Ultrasound therapy combined with standard cream + conventional moisturizing and sunscreen
  Arms: Control group

SUMMARY:
A Prospective, Single-center, Single-blind, Randomized split-face, controlled trial will be conducted. The goal of this clinical trial is to evaluate the efficacy and satisfaction of ultrasound therapy combined with SkinCeuticals A.G.E in improving facial aging, and to explore the medical value of ultrasound therapy combined with SkinCeuticals A.G.E. Participants will be treated with ultrasound combined with SkinCeuticals A.G.E on one randomized side face and ultrasound combined with standard cream on the other side.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 18-65 years inclusive;
2. The subject 's facial skin is rough, flaccid, and lack of elasticity;
3. Subjects with multiple facial fine lines (perioral/periocular/forehead, etc.), decree lines or puppet lines area with static fine lines trend, the lower part showed signs of loosening;
4. Subjects who have consistent facial skin status on both sides and plan to receive ultrasound therapy;
5. Subjects are willing to follow the requirements of the study protocol and complete the corresponding procedures;
6. Subjects understand the nature of the study and sign the informed consent form (ICF).

Exclusion Criteria:

1. Subjects with contraindications to ultrasound treatment (such as malignant tumor, acute systemic infection, severe heart disease, bleeding tendency, etc.) or contraindications to A.G.E use (or allergic to other skin care components);
2. Subjects with facial skin diseases, infection, inflammation or allergic constitution that may affect the judgment of the test results;
3. Subjects with hypertrophic scar or scar constitution;
4. Receiving treatment of tightening medical treatment program (Thermage/Fotona 4D/ultrasound/microneedle, etc.) or planning to receive other tightening medical treatment program and drugs during this treatment in the past 3 months;
5. Patients who have oral or topical cosmetic products that may affect the test results within the past 2 weeks;
6. Subjects who have participated in drug clinical trials or other trials within the past 30 days (or are participating in), or have used drugs affecting the test results within 1 week;
7. Female subjects who are pregnant, lactating or plan to become pregnant;
8. Other subjects who are not suitable for participating in this study as assessed by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Global aesthetic improvement scale （GAIS） score | at day 90 after procedure
  Investigator Satisfaction Assessment Form. Scoring criteria: 5 (very much improved), 4 (marked improvement), 3 (improved), 2 (no change), or 1 (worse).

SECONDARY OUTCOMES:
Change from baseline in fine lines score | at 30, 60, 90, 180 days after procedure
  Skin Parameter Assessment Form. Fine lines: Grading was performed on a Griffith 's scale (10-point scale) with different scores representing: 0 (no fine lines/wrinkles, skin completely smooth and no wrinkles); 1-3 (mild, few fine lines and wrinkles, and distant intervals within the treatment area); 4-6 (moderate, moderate number of fine lines/wrinkles within the treatment area and close to each other); and 7-9 (severe, dense clusters of fine lines/wrinkles within the treatment area). Fine lines status should be evaluated by an independent investigator.
Relative change from baseline in skin elasticity | at 30, 60, 90, 180 days after procedure
Relative change from baseline in dermal thickness | at 30, 60, 90, 180 days after procedure
Relative change in transepidermal water loss(TEWL) from baseline | at 30, 60, 90, 180 days after procedure
Investigator satisfaction assessment | at 30, 60, 90, 180 days after surgery
  Investigator Satisfaction Assessment Form. Questions included: 1. Integrated skincare effect of ultrasonic program. 2, Feeling overall improvement of facial wrinkles after using the product. 3, Feeling that the elasticity of facial skin is improved after using the product. 4, Feeling that facial skin fullness improved after using the product. 5. Feeling that the skin moisture is improved after using the product. Satisfaction ratings were divided into: 1: very dissatisfied, 2: dissatisfied, 3: fair, 4: satisfied, and 5: very satisfied, and the proportion of people in each rating was statistically summarized
Subject satisfaction evaluation | at 30, 60, 90, 180 days after procedure
  Subject Satisfaction Assessment Form. Questions included: 1. Integrated skincare effect of ultrasonic program. 2, Feeling overall improvement of facial wrinkles after using the product. 3, Feeling that the elasticity of facial skin is improved after using the product. 4, Feeling that facial skin fullness improved after using the product. 5. Feeling that the skin moisture is improved after using the product. Satisfaction ratings were divided into: 1: very dissatisfied, 2: dissatisfied, 3: fair, 4: satisfied, and 5: very satisfied, and the proportion of people in each rating was statistically summarized
Global aesthetic improvement scale （GAIS） score | at day 30,60,180 after procedure
  Investigator Satisfaction Assessment Form. Scoring criteria: 5 (very much improved), 4 (marked improvement), 3 (improved), 2 (no change), or 1 (worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Hang Zhou YesSkin Hospital, Hangzhou, China

REFERENCES:
- [Derived] Jiang X, Peng S, Chen Y, Nan Y, Song W. A Randomized, Investigator-Blinded, Split-Face, Controlled Trial Evaluating the Efficacy and Satisfaction of a Topical Product Containing Blueberry Extract and Pro-Xylane Combined With Micro-Focused Ultrasound for Anti-aging. J Cosmet Dermatol. 2025 Jul;24(7):e70281. doi: 10.1111/jocd.70281. PMID 40635529